CLINICAL TRIAL: NCT00809926
Title: An 8-week Randomized, Double-Blind, Parallel Group, Multi-Center, Active Controlled Study to Evaluate the Efficacy and Safety of Valsartan Administered in Combination With Aliskiren (160/150 mg, 320/300 mg) Versus Valsartan Alone (160 mg, 320 mg) in Patients With Stage 2 Hypertension
Brief Title: 8 Weeks Study to Evaluate the Efficacy and Safety of Valsartan in Combination With Aliskiren Compared to Valsartan Alone in Patients With Stage 2 Hypertension
Acronym: VANTAGE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSPV100AUS01
Record Dates: First submitted 2008-12-16; First posted 2008-12-17 (Estimated); Results first posted 2011-05-02 (Estimated); Last update posted 2011-05-02 (Estimated); Status verified 2011-03

CONDITIONS: Stage 2 Hypertension
Keywords: Hypertension, aliskiren and valsartan
MeSH Terms: conditions — Hypertension | interventions — Valsartan; aliskiren

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Valsartan/aliskiren (Experimental)
  Interventions: Drug: Valsartan/aliskiren
- Valsartan (Active Comparator)
  Interventions: Drug: Valsartan

INTERVENTIONS:
Drug: Valsartan/aliskiren — Valsartan/aliskiren (160/150mg) for 2 weeks followed by forced titration to valsartan/aliskiren (320/300mg) for the remaining 6 weeks
  Arms: Valsartan/aliskiren
Drug: Valsartan — Valsartan (160mg) for 2 weeks followed by forced titration to Valsartan (320mg) for the remaining 6 weeks
  Arms: Valsartan

SUMMARY:
To evaluate the efficacy and safety of the valsartan/aliskiren combination compared to valsartan alone in patients with Stage 2 hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are eligible and able to participate in the study, and who give written informed consent before any assessment is performed.
* Men or women 18 years and older.
* Patients with Stage 2 systolic hypertension; defined as having a MSSBP ≥160 mmHg and <180 mmHg at Visit 5 (randomization).

Exclusion Criteria:

* Use of aliskiren or participation in a clinical trial that had aliskiren as treatment within 30 days of Visit 1.
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test (>5 mIU/ml).
* Women of child-bearing potential (WOCBP), defined as all women physiologically capable of becoming pregnant, including women whose career, lifestyle, or sexual orientation precludes intercourse with a male partner and women whose partners have been sterilized by vasectomy or other means, UNLESS they meet the following definition of post-menopausal: 12 months of natural (spontaneous) amenorrhea or 6 months of spontaneous amenorrhea with serum FSH levels >40 mIU/m or 6 weeks post surgical bilateral oophorectomy with or without hysterectomy OR are using one or more of the following acceptable methods of contraception: surgical sterilization (e.g., bilateral tubal ligation), hormonal contraception (implantable, patch, oral), and double-barrier methods. Reliable contraception should be maintained throughout the study and for 7 days after study drug discontinuation.
* Severe hypertension (an office cuff MSDBP ≥110 mmHg and/or MSSBP ≥180 mmHg).
* Refractory hypertension, defined as unresponsive to triple drug therapy at the maximum dose of each drug, one of which must be a diuretic, and not at blood pressure goal (140/90 mmHg).
* Patients treated with more than 3 antihypertensive medications (each component of a combination drug counts individually).
* History or evidence of a secondary form of hypertension.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 451 (Actual)
Dates: Start 2009-01; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Chair — Novartis
Locations (1):
- Sites in USA, East Hanover, New Jersey, United States

REFERENCES:
- [Derived] Flack JM, Yadao AM, Purkayastha D, Samuel R, White WB. Comparison of the effects of aliskiren/valsartan in combination versus valsartan alone in patients with stage 2 hypertension. J Am Soc Hypertens. 2012 Mar-Apr;6(2):142-51. doi: 10.1016/j.jash.2011.11.004. Epub 2012 Feb 9. PMID 22321963

RESULTS

PARTICIPANT FLOW:
Groups:
- Valsartan/Aliskiren: For the first 2 weeks patients received Valsartan/aliskiren (160/150mg). For the remaining 6 weeks, all patients received Valsartan/aliskiren 320/300mg (forced titration).
- Valsartan: For the first 2 weeks patients received Valsartan 160 mg. For the remaining 6 weeks, all patients received Valsartan 320 mg (forced titration).
Period: Overall Study
Arm/Group | Valsartan/Aliskiren | Valsartan
Started | 232 | 219
Completed | 201 | 196
Not Completed | 31 | 23
Not completed — Adverse Event | 18 | 10
Not completed — Unsatisfactory therapeutic effect | 3 | 3
Not completed — Patient withdrew consent | 8 | 6
Not completed — Lost to Follow-up | 2 | 1
Not completed — Administrative Problems | 0 | 1
Not completed — Protocol deviation | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Valsartan/Aliskiren | Valsartan | Total
Number analyzed (Participants) | 232 | 219 | 451
Age Continuous [Mean (Standard Deviation); unit: years] | 57.5 (11.1) | 56.7 (11.0) | 57.1 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107 | 116 | 223
  Male | 125 | 103 | 228

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Sitting Systolic Blood Pressure (MSSBP) at Week 8
Description: To compare the change from baseline in MSSBP after 8 weeks of treatment with a valsartan and aliskiren treatment regimen (160/150 mg, 320/300 mg) versus a valsartan treatment regimen (160 mg, 320 mg) in patients with Stage 2 Hypertension.
Time Frame: Baseline to Week 8
Population: Intent-to-treat (ITT) population consisted of all randomized patients who received at least 1 dose of study drug and had valid baseline and 1 valid post-baseline assessment of an efficacy variable. The last-observation-carried-forward (LOCF) method was used for replacing the missing values of the post-baseline assessments for ITT analysis at wk 8.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Valsartan/Aliskiren | Valsartan
Number analyzed (Participants) | 230 | 217
mm Hg
  Baseline | 164.8 (4.54) | 166.2 (5.23)
  Week 8 | 142.3 (17.01) | 145.6 (17.55)
  Change from Baseline to Week 8 | -22.5 (16.04) | -20.6 (16.25)
Statistical Analysis 1: Comparison: Valsartan/Aliskiren vs Valsartan; Test type: Superiority or Other; p = 0.295, ANCOVA; Least Square Mean Difference = -1.6, 95% CI 2-sided [-4.61 to 1.40]

2. Secondary Outcome: Change From Baseline in Mean Sitting Diastolic Blood Pressure (MSDBP) at Week 8
Description: To compare the change in MSDBP after 8 weeks of treatment with a valsartan and aliskiren treatment regimen (160/150 mg, 320/300 mg) versus a valsartan (160 mg, 320 mg) treatment regimen in patients with Stage 2 Hypertension.
Time Frame: Baseline to Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Valsartan/Aliskiren | Valsartan
Number analyzed (Participants) | 230 | 217
mm Hg
  Baseline | 93.9 (8.22) | 94.8 (8.68)
  Week 8 | 85.7 (10.94) | 86.4 (10.34)
  Change from Baseline to Week 8 | -8.2 (9.77) | -8.3 (9.49)
Statistical Analysis 1: Comparison: Valsartan/Aliskiren vs Valsartan; Test type: Superiority or Other; p = 0.790, ANCOVA; Least Square Mean Difference = -0.2, 95% CI 2-sided [-1.93 to 1.47]

3. Secondary Outcome: Percentage of Patients Achieving Blood Pressure Control (Defined as Patients Achieving a MSSBP <140 mmHg and MSDBP <90 mmHg) at Week 8
Description: To evaluate the percentage of patients achieving blood pressure control (defined as patients achieving a MSSBP <140 mmHg and MSDBP <90 mmHg) at week 8 following treatment with a valsartan and aliskiren treatment regimen (160/150 mg, 320/300 mg) versus a valsartan treatment regimen (160 mg, 320 mg) in patients with Stage 2 Hypertension.
Time Frame: At Week 8
Population: The intent-to-treat (ITT) population consisted of all randomized patients who received at least one dose of study medication and had valid baseline and at least one valid post-baseline assessment of an efficacy variable.
Measure: Number; unit: percentage of patients
Arm/Group | Valsartan/Aliskiren | Valsartan
Number analyzed (Participants) | 230 | 217
percentage of patients | 44.3 | 36.2
Statistical Analysis 1: Comparison: Valsartan/Aliskiren vs Valsartan; Test type: Superiority or Other; p = 0.101, Cochran-Mantel-Haenszel; Difference = 8.1, 95% CI 2-sided [-1.56 to 17.67]

4. Secondary Outcome: Percentage of Responders (Defined as Patients With MSSBP <140 mmHg or a Decrease From Baseline ≥20 mmHg) at Week 8
Description: To compare the percentage of responders (defined as patients with MSSBP <140 mmHg or a decrease from baseline ≥20 mmHg) at week 8 following treatment with a valsartan and aliskiren treatment regimen (160/150 mg, 320/300 mg) versus a valsartan treatment regimen (160 mg, 320 mg) in patients with Stage 2 Hypertension.
Time Frame: At Week 8
Population: as for outcome 3
Measure: Number; unit: percentage of responders
Arm/Group | Valsartan/Aliskiren | Valsartan
Number analyzed (Participants) | 230 | 217
percentage of responders | 64.7 | 53.1
Statistical Analysis 1: Comparison: Valsartan/Aliskiren vs Valsartan; Test type: Superiority or Other; p = 0.018, Cochran-Mantel-Haenszel; Difference = 11.6, 95% CI 2-sided [2.00 to 21.33]

5. Secondary Outcome: Mean Change From Baseline in Plasma Renin Activity (PRA) at Week 8
Description: To assess the change from baseline in PRA after 8 weeks of treatment with a valsartan and aliskiren treatment regimen (160/150 mg, 320/300 mg) versus a valsartan treatment regimen (160 mg, 320 mg) in patients with Stage 2 Hypertension.
Time Frame: Baseline to Week 8
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/mL/h
Arm/Group | Valsartan/Aliskiren | Valsartan
Number analyzed (Participants) | 230 | 217
ng/mL/h
  Baseline | 0.992 (1.290) | 0.831 (0.854)
  Week 8 | 0.436 (0.659) | 2.450 (3.73)
  Change from Baseline to Week 8 | -0.540 (1.285) | 1.577 (3.528)

6. Secondary Outcome: Mean Change From Baseline in Plasma Renin Concentration (PRC) at Week 8
Description: To assess the change from baseline in PRC after 8 weeks of treatment with a valsartan and aliskiren treatment regimen (160/150 mg, 320/300 mg) versus a valsartan treatment regimen (160 mg, 320 mg) in patients with Stage 2 Hypertension.
Time Frame: Baseline to Week 8
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Valsartan/Aliskiren | Valsartan
Number analyzed (Participants) | 230 | 217
ng/L
  Baseline | 8.286 (10.893) | 8.065 (14.932)
  Week 8 | 142.833 (293.228) | 20.089 (31.771)
  Change from Baseline to Week 8 | 135.515 (296.758) | 11.988 (32.679)

7. Other Pre Specified Outcome: Completers Analysis for Change From Baseline in MSSBP at Week 8
Description: To evaluate the change from baseline in MSSBP (mmHg) at Week 8; primary efficacy variable at primary time point in ITT population - patients who completed the double-blind treatment period.
Time Frame: Baseline to week 8
Population: The analysis included ITT patients who completed the double-blind treatment period [those patients with a final observation at week 8, also known as observed cases (OC)]. This analysis differed from the ITT-LOCF analysis, in that it did not include patients who discontinued from the trial prematurely.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Valsartan/Aliskiren | Valsartan
Number analyzed (Participants) | 201 | 196
mm Hg
  Baseline | 164.8 (4.54) | 166.2 (5.23)
  Week 8 | 140.9 (15.74) | 145.9 (16.89)
  Change from Baseline to Week 8 | -24.0 (14.70) | -20.3 (15.49)
Statistical Analysis 1: Comparison: Valsartan/Aliskiren vs Valsartan; Test type: Superiority or Other; p = 0.028, ANCOVA; Least Square Mean Difference = -3.4, 95% CI 2-sided [-6.34 to -0.37]

8. Other Pre Specified Outcome: Longitudinal Repeated Measure Analysis for Change in MSSBP From Baseline Through Week 8
Description: To evaluate the change from baseline in MSSBP (mmHg) after 8 weeks; primary efficacy variable (ITT population) using Longitudinal analysis (A repeated measures analysis where assessments over time are considered , as opposed to looking at a single point in time.)
Time Frame: Baseline through week 8
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Valsartan/Aliskiren | Valsartan
Number analyzed (Participants) | 230 | 217
mm Hg | -23.2 (1.04) | -20.1 (1.08)
Statistical Analysis 1: Comparison: Valsartan/Aliskiren vs Valsartan; Test type: Superiority or Other; p = 0.040, GENMOD; Based on a generalized estimating equations using SAS procedure GENMOD; Least Square Mean Difference = -3.1, 95% CI 2-sided [-6.02 to -0.14]

9. Other Pre Specified Outcome: Change From Baseline in Mean Ambulatory Systolic Blood Pressure (MASBP).
Description: To evaluate 24-hour ambulatory systolic blood pressure measurements in a subset of patients after 8 weeks of treatment with the combination of valsartan and aliskiren versus valsartan monotherapy in patients with stage 2 hypertension.
Time Frame: Baseline to week 8
Population: Patients who were willing to participate in the Ambulatory Blood Pressure Monitoring (ABPM) substudy and who met the study inclusion and exclusion criteria for randomization.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Valsartan/Aliskiren | Valsartan
Number analyzed (Participants) | 58 | 53
mm Hg
  Baseline | 146.1 (9.14) | 143.5 (14.10)
  Week 8 | 130.3 (13.41) | 137.6 (17.11)
  Change from Baseline to Week 8 | -15.8 (11.42) | -6.0 (13.34)
Statistical Analysis 1: Comparison: Valsartan/Aliskiren vs Valsartan; Test type: Superiority or Other; p = 0.004, ANCOVA; Least Square Mean Difference = -8.7, 95% CI 2-sided [-14.38 to -2.93]

10. Other Pre Specified Outcome: Change From Baseline in Mean Ambulatory Diastolic Blood Pressure (MADBP)
Description: To evaluate 24-hour ambulatory diastolic blood pressure measurements in a subset of patients after 8 weeks of treatment with the combination of valsartan and aliskiren versus valsartan monotherapy in patients with stage 2 hypertension.
Time Frame: Baseline to week 8
Population: Patients who were willing to participate in the ABPM substudy and who met the study inclusion and exclusion criteria for randomization.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Valsartan/Aliskiren | Valsartan
Number analyzed (Participants) | 58 | 53
mm Hg
  Baseline | 87.9 (7.28) | 85.7 (9.26)
  Week 8 | 78.2 (9.44) | 81.7 (10.11)
  Change from Baseline to Week 8 | -9.7 (7.02) | -4.0 (8.09)
Statistical Analysis 1: Comparison: Valsartan/Aliskiren vs Valsartan; Test type: Superiority or Other; p = 0.006, ANCOVA; Least Square Mean Difference = -4.9, 95% CI 2-sided [-8.37 to -1.42]

ADVERSE EVENTS:
Time Frame: Baseline through week 8
Groups:
- Valsartan/ Aliskiren: Valsartan/aliskiren (160/150mg) for 2 weeks followed by forced titration to valsartan/aliskiren (320/300mg) for the remaining 6 weeks
- Valsartan: Valsartan (160mg) for 2weeks followed by forced titration toValsartan (320mg) for the remaining 6 weeks
Arm/Group | Valsartan/ Aliskiren | Valsartan
Serious Adverse Events (participants affected / at risk) | 5/232 | 3/219
Other Adverse Events (participants affected / at risk) | 14/232 | 15/219
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Valsartan/ Aliskiren (N=232) | Valsartan (N=219)
Lymphocytosis (Blood and lymphatic system disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Chest discomfort (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 2 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Anaesthesia (Nervous system disorders) | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1
Conversion disorder (Psychiatric disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Valsartan/ Aliskiren (N=232) | Valsartan (N=219)
Headache (Nervous system disorders) | 14 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.